CLINICAL TRIAL: NCT00115609
Title: Pilot Trial Evaluating Once Daily Triple Combination Antiretroviral Therapy With Tenofovir-Emtricitabine and Efavirenz in HIV-1 Infected Patients With Mycobacterium Tuberculosis Infection ANRS129 BKVIR
Brief Title: Efficacy of Tenofovir-Emtricitabine and Efavirenz in HIV Infected Patients With Tuberculosis (ANRS129)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-002470-30; ANRS129 BKVIR
Record Dates: First submitted 2005-06-23; First posted 2005-06-24 (Estimated); Last update posted 2011-12-22 (Estimated); Status verified 2011-12

CONDITIONS: HIV Infections; Tuberculosis
Keywords: HIV infections; tuberculosis; tuberculosis agents; Anti HIV agents; Treatment Naive
MeSH Terms: conditions — HIV Infections; Tuberculosis | interventions — efavirenz; Tenofovir; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: efavirenz — 800mg for patients treated by rifampicine 600mg for other patients
  Other Names: Sustiva
Drug: tenofovir DF — 300mg once a day
  Other Names: Viread
Drug: emtricitabine — one pill of 200mg once a day
  Other Names: Emtriva/FTC

SUMMARY:
Successful therapy of both tuberculosis and HIV disease share similar problems: pill burden, drug interaction, adherence challenge and toxicity. This study will test the efficacy and safety of a once daily antiretroviral regimen in HIV-tuberculosis coinfected patients.

DETAILED DESCRIPTION:
The proposed research consists of conducting a pilot trial "BKVIR" designed to answer the question of whether once daily tenofovir-emtricitabine-efavirenz triple-agent therapy is effective and well tolerated when it must be initiated within three months after initiation of a three-agent or four-agent tuberculostatic therapy in antiretroviral-naive HIV-infected patients. As the proposed pilot trial comprises the initiation of antiretroviral therapy during the three months following the initiation of tuberculostatic therapy, we propose to set up systematic, continuous registration of HIV-infected patients with a diagnosis of tuberculosis in participating centers during the study period in order to evaluate their eligibility for inclusion in the pilot trial. The initial declaration phase in the register, in addition to facilitating inclusions in the pilot trial, should also allow: 1) a better understanding of the reasons for non-inclusion in the trial, allowing the eligibility criteria to be adjusted if necessary during the trial; and 2) to describe the antiretroviral therapies used during co-infection and their time of initiation in relation to tuberculostatic therapy.

This research is expected to contribute to an updating of the treatment guidelines in the context of tuberculosis in HIV-infected patients. The data collected will constitute a unique database on this issue not only in France, but also internationally, which will also be useful to optimize management strategies of these two diseases in developing countries.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years
* Infected by HIV-1
* Naive to antiretroviral therapy
* Presenting an indication to start antiretroviral therapy (according to the recommendations of the Delfraissy 2004 report)
* Histologically or microbiologically confirmed tuberculosis
* Receiving tuberculostatic therapy for less than three months

Exclusion Criteria:

* Isolated HIV-2 infection
* Neoplasm treated by chemotherapy and/or radiotherapy
* Pregnancy or plans for pregnancy
* Breastfeeding
* Contraindication to one of the antiretroviral drugs
* Atypical mycobacterial infection
* Hemoglobin below 8 g/dL
* Neutrophils below 750/mm3
* Platelets below 50,000/mm3
* Creatinine clearance below 60 ml/min
* Alkaline phosphatase, ASAT, ALAT or bilirubin over 3 times the upper limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-01; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
treatment success rate at week 48 (W48) | W48

SECONDARY OUTCOMES:
course of plasma HIV-1 RNA between W0 and W48 | W48
tuberculosis cure rate | W48
safety of trial treatments (number of events, description, time to onset, metabolic disorders, immune restoration syndrome) | W48
frequency of treatment changes or discontinuations | W48
clinical progression of HIV infection | W48
course of CD4 and CD8 T lymphocytes | W48
study of resistance in the case of virological failure | W48
study of compliance and quality of life | W48
pharmacokinetic study of tuberculostatic agents | W02,W08,W12, W24
effect of treatment on hepatitis B viral replication | W48

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Lortholary, MD, Principal Investigator — Hopital Necker-Enfants malades; Geneviève Chêne, MD, Study Director — INSERM U593
Locations (1):
- Service des maladies Infectieuses et tropicales Hopital Necker-Enfants Malades, Paris, France

REFERENCES:
- See also: Related Info — http://www.anrs.fr